CLINICAL TRIAL: NCT06464237
Title: Metacognitive Intervention in Youth With Oncological Disease - the Mio Study
Acronym: Mio
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BASEC2023-01196
Record Dates: First submitted 2024-06-12; First posted 2024-06-18 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Cancer
Keywords: Metacognition; Pediatric cancer; Neurorehabilitation; Cognitive training; Physical training; Adolescents with cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training group (Active Comparator): Training with Mio-App for 5 weeks, three times per week.
  Interventions: Behavioral: Mio-App
- Control group (No Intervention): Waiting control group. Participants may use the Mio-App after completion of the last follow-up assessment.

INTERVENTIONS:
Behavioral: Mio-App — The Mio-App aims to increase metacognitive knowledge, teaches mnemonic skills, trains the working memory capacity and motor skills to reduce cognitive and physical long-term sequelae after cancer during adolescence.
  Other Names: Mio-Training
  Arms: Training group

SUMMARY:
The aim of the Mio-Study is to address the current lack of effective treatment options to reduce cognitive and physical long-term problems in children and adolescents with cancer. Through the use of the Mio-App, cognitive and physical development will be strengthened and metacognitive thinking and awareness will increase.

The Mio-App for children and adolescence with cancer will include a combination of cognitive and physical training tasks and prospective as well as retrospective metacognitive questions. In a randomized controlled trial, the App will be analysed for its efficacy on metacognitive thinking and executive functions. In particular, the investigators are interested in factors that affect the efficacy of the training program such as compliance, age, sex or the presence of fatigue. This study will give insight into the role of metacognition in cognitive and physical performance and will foster the development of children and adolescents with cancer in the long-term.

DETAILED DESCRIPTION:
In the Mio-Study, the investigators are developing a training app at the interface between neuropsychology and sports science - the Mio-training. The aim of the Mio-training is to strengthen the cognitive and motor development of children and adolescents after cancer in the long-term. The App contains a combination of cognitive and physical training tasks and metacognitive questions to promote knowledge and awareness of one's own thinking. In order to counteract the shortage of skilled workers and the increasing specialization of individual specialist areas, solutions are needed that can be implemented without a lot of staff. From today's perspective, there are hardly any trainings for children and adolescents that show long-term effects on cognitive and motor development and can also be transferred to non-trained tasks in school and everyday life.

The investigators are testing the effectiveness of the Mio-training in a randomized clinical trial (RCT) and expect a strengthening of metacognition and core cognitive functions (i.e. executive functions). The Mio-Study will provide information about the role of metacognition in cognitive and physical performance and, ideally, provide evidence for a novel, interdisciplinary rehabilitation strategy for children and adolescents after cancer.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent as documented by signature (see Informed Consent Form) of participants and / or parents / legal guardians
* Age 8-16 years
* A diagnosis of cancer either with or without CNS involvement. The participant will be included between 3 months before to 10 years after termination of treatment.
* Treatment of cancer including either radiation, chemotherapy and/ or surgical tumor removal
* German or French speaking

Exclusion Criteria:

* Any other instable neurological condition (e.g. epilepsy)
* A severe psychiatric disease (e.g., eating disorder) or severe learning disability
* Known or suspected non-compliance
* Drug or alcohol abuse
* Inability to follow the procedures of the study, e.g. due to language problems
* Enrolment of the investigator, his/her family members, employees and other dependent persons

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Junior Metacognitive Awareness Inventory | At baseline; immediately (up to 1 week) after the training or waiting period; at 3-months follow-up
  Total score of the Junior Metacognitive Awareness Inventory over the three timepoints (baseline, immediate followup & 3-months follow-up). Raw values ranging 18-90. Higher scores mean better outcome.

SECONDARY OUTCOMES:
Wechsler Intelligence Scale For Children: 5th Ed (WISC-V) | At baseline; immediately (up to 1 week) after the training or waiting period.
  Indices ranging from 0 to 155. Higher scores mean better outcome.
Color-Word Interference Test | At baseline; immediately (up to 1 week) after the training or waiting period.
  Scaled Scores ranging from 1 to 19. Higher scores mean better outcome.
Tower of Hanoi (D-KEFS) | At baseline; immediately (up to 1 week) after the training or waiting period.
  Scaled Scores ranging from 1 to 19. Higher scores mean better outcome.
Verbal learning and memory test (VLMT) | At baseline; immediately (up to 1 week) after the training or waiting period.
  Percentile ranks ranging from 0-100. Higher scores mean better outcome.
Pattern learning (Basic-MLT) | At baseline; immediately (up to 1 week) after the training or waiting period.
  Percentile ranks ranging from 0-100. Higher scores mean better outcome.
German Motor Performance Test (DMT) | At baseline; immediately (up to 1 week) after the training or waiting period.
  Percentile ranks ranging from 0-100. Higher scores mean better outcome.
Behaviour Rating Inventory of Executive Function | At baseline; immediately (up to 1 week) after the training or waiting period; at 3-months follow-up.
  Percentile ranks ranging from 0-100. Higher scores mean better outcome.

OTHER OUTCOMES:
Physical Self-Description Questionnaire (PSDQ-S) | At baseline; immediately (up to 1 week) after the training or waiting period; at 3-months follow-up.
  Short version, Likert scale ranging from 1 to 6. Higher scores mean better outcome.
Questionnaire for the Assessment of Resources and Competencies in Childhood and Adolescence (FRKJ) | At baseline; immediately (up to 1 week) after the training or waiting period; at 3-months follow-up.
  Stanine rank from 1-9. Higher score mean better outcome.
Pediatric quality of life multidimensional fatigue scale (PedsQL-MFS) | At baseline; immediately (up to 1 week) after the training or waiting period; at 3-months follow-up.
  5-point Likert scale ranging from 0 to 4. Higher scores mean better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Regula Everts, Prof. Dr., Principal Investigator — Division of Neuropaediatrics, Development and Rehabilitation, Department of Paediatrics, Inselspital, Bern University Hospital, University of Bern, Switzerland
Locations (1):
- Insespital, University Hospital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No
Data can be shared upon reasonable request

REFERENCES:
- See also: Link to Mio-Study — https://kinderklinik.insel.ch/de/lehre-und-forschung/forschung/forschung-nach-fachgebiet/neuropaediatrie/research-projects/mio-studie